CLINICAL TRIAL: NCT05529940
Title: Efficacy of Perioperative Versus Adjuvant FOLFIRINOX in Resectable Pancreatic Cancer: an International Multicenter Randomized Controlled Trial (NeoFOL-R Trial)
Brief Title: NeoFOL-R Trial (Perioperative Versus Adjuvnat FOLFIRINOX in Resectable Pancreatic Cancer)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other); SMG-SNU Boramae Medical Center (Other); Gangnam Severance Hospital (Other); Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Jin-Young Jang, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-2211-115-1380
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Resectable Pancreatic Cancer; Neoadjuvant Chemotherapy; Effects of Chemotherapy
MeSH Terms: interventions — folfirinox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neoadjuvant FOLFIRINOX (Experimental): 6 cycles of neoadjuvant mFOLFIRINOX followed by surgical resection and 6 cycles of adjuvant mFOLFIRINOX
  Interventions: Drug: Folfirinox
- Upfront Surgery (Active Comparator): surgical resection followed by 12 cycles of adjuvant mFOLFIRINOX
  Interventions: Drug: Folfirinox

INTERVENTIONS:
Drug: Folfirinox — The primary aim of this trial was to investigate whether six cycles of preoperative mFOLFIRINOX followed by six cycles of postoperative mFOLFIRINOX improved the overall survival rate by intention-to-treat compared to surgery followed by 12 cycles of postoperative mFOLFIRINOX.

SUMMARY:
Rationale: Adjuvant chemotherapy after surgery significantly improved the survival of PC patients, but there is a problem that only about 50% of patients start adjuvant chemotherapy after pancreatectomy. Neoadjuvant chemotherapy might control potential metastatic lesion which are not being detected in early diseases status and improve the R0 resection rate. In addition, it prevents futile surgery by selecting patients with rapid progression of disease. Furthermore, compared to chemotherapy administered after surgery, more patients can complete the planned chemotherapy schedule in neoadjuvant setting. Asians differ from Westerners not only in racial differences, but also in average size and body surface area. Accordingly, there is an urgent need for clinical studies on the dose, toxicity, dosing cycle, and efficacy of anticancer drugs that reflect actual clinical trials in Asian countries for Asians. There are still few studies worldwide that prospectively explored the efficacy of neoadjuvant chemotherapy in resectable PC and the administration of neoadjuvant therapy in resectable PC depends on individual clinical judgment. Therefore, systematic and prospective clinical trials are essential to standardize treatment protocol in resectable PC.

Obective: To investigate whether 6 cycles of preoperative mFOLFIRINOX - surgery - 6 cycles of postoperative mFOLFIRINOX improves overall survival by intention-to-treat compared to surgery followed by 12 cycles of postoperative mFOLFIRINOX.

Study design: open-label, multicenter, randomized, phase 3 clinical trial Study population: Patients with resectable pancreatic cancer and ECOG performance 0 or 1.

Intervention:

Invervention arm : 6 cycles of neoadjuvant mFOLFIRINOX followed by surgical resection and 6 cycles of adjuvant mFOLFIRINOX Comparator arm : surgical resection followed by 12 cycles of adjuvant mFOLFIRINOX Primary endpoint: 2-year overall survival rate by intention-to-treat

ELIGIBILITY:
Inclusion Criteria:

- A. Age: 19 to 80 years old B. Patients with a score of 0 - 1 (ECOG) when selecting a study subject C. Pancreatic ductal adenocarcinoma diagnosed by histological examination (histologic or cytopathological) D. Patients evaluated as resectable pancreatic cancer in preoperative imaging as follows (NCCN guidelines for pancreatic adenocarcinoma version 2.2021)

* No arterial tumor contact (celiac asix, superior mesenteric artery, or common hepatic artery).
* No tumor contact with the superior mesenteric vein or portal vein or ≤ 180°contact without vein contour irregularity.

E. No distant metastases on preoperative imaging F. Patients with adequate organ function

1. Bone marrow function: WBC 3,000/mm3 or more or ANC 1,500/mm3 or more, platelet ≥ 100K/mm3
2. Liver function: Bilirubin ≤ 3 x upper normal limit (≤5.0 mg/dL), AST/ALT ≤ 5 x upper normal limit (<200 IU/L)
3. Renal function (Cr clearance ≥ 60 mL/min) or (Cr < 1.5 x upper normal limit) G. Persons physically capable of undergoing surgery H. Those who consented to the clinical trial I. Women of childbearing potential must have a negative serum pregnancy test within one week before starting the intervention drug. Men and women of childbearing potential must use effective contraception from screening through six months after the last dose.

Exclusion Criteria:

- Patients who met any of the following criteria are not eligible to participate in this study.

A. Those evaluated as borderline resectable or locally advanced pancreatic cancer in preoperative imaging examination (The resectability assessment depends on the presence of major vessel invasion, while invasion of adjacent organs is excluded from the criteria) B. Patients with a history of previous pancreatic surgery C. Patients with a history of previous chemotherapy or radiation therapy for pancreatic cancer D. Patients with distant metastases or recurrent pancreatic cancer E. Pancreatic body or tail cancer requiring combined resection of adjacent organs (stomach or kidney) (except for the adrenal gland) F. Patients within five years of diagnosis of other organ malignancies (with the exception of adequately treated non-melanoma skin cancer and carcinoma in situ without evidence of disease) G. Pregnant and lactating women H. Serious concomitant systemic disorders, including active or ongoing systemic infections, symptomatic congestive heart failure, unstable angina, clinically significant cardiac arrhythmias, psychiatric disorders, or uncontrolled comorbid conditions that may limit compliance with study requirements, or any medical condition that, at the discretion of the investigator, could compromise patient safety, interfere with the assessment of safety and efficacy, or hinder participation in the clinical trial.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 609 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
2-year survival rate | 2 years
  The primary objective of this trial is to investigate whether 6 cycles of preoperative mFOLFIRINOX - surgery - 6 cycles of postoperative mFOLFIRINOX improves overall survival by intention-to-treat compared to surgery followed by 12 cycles of postoperative mFOLFIRINOX.

SECONDARY OUTCOMES:
Overall survival | 5 years
  Defined as the time from the date of randomization to the date of death from any cause. Patients who were not reported dead at the time of analysis were censored on the last day they were known to be alive.
Disease free survival | 3 years
  Defined as the time between the date of randomization and the occurrence of distant metastases, locoregional progression, or death from any cause. Patients who were alive and free of these events at the last follow-up would be censored.
Resection rate | 3 years
  Referred to the proportion of patients who underwent curative resection
R0 resection rate | 3 years
  Referred to the proportion of patients with microscopically negative resection margins due to the pathological examinations after the surgery. In this case, R0 indicated that no tumor was observed within 0 mm from the margins of resection.
Local recurrence rate | 3 years
  Local recurrence is defined as recurrence in the pancreatic resection margin, residual pancreas, and regional lymph nodes, and distant metastasis is defined as recurrence in a distant organ. The local recurrence and distant metastasis rates are defined as the percentage of patients who had recurrence after the surgical resection.
Recurrence rate | 2 year
  The proportion of patients who experienced recurrence within two years from the date of surgery.
Response rate in neoadjuvant setting | 3 years
  Defined as the percentage of patients who showed complete response, partial response, and stable disease after three or six cycles of scheduled chemotherapy. The evaluation is based on RECIST v.1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Wooil Kwon, Study Director — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Department of Internal Medicine, Seoul St. Mary's Hospital, Catholic University College of Medicine, Seoul
  - Department of Surgery, Seoul National University College of Medicine, Seoul

IPD SHARING:
Plan to Share IPD: No